CLINICAL TRIAL: NCT07018635
Title: An Open-Label Study to Assess the Effect of Itraconazole, Rifampin, and Acid-Reducing Agents on INCB161734 Pharmacokinetics When Administered Orally in Healthy Participants
Brief Title: A Study to Assess the Effect of Itraconazole, Rifampin, and Acid-Reducing Agents on INCB161734 Pharmacokinetics When Administered Orally in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INCB161734-103
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants
Keywords: INCB161734
MeSH Terms: interventions — Itraconazole; Rifampin; Esomeprazole; Famotidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): INCB161734 and itraconazole will be administered at protocol defined doses.
  Interventions: Drug: INCB161734; Drug: Itraconazole
- Cohort 2 (Experimental): INCB161734 and rifampin will be administered at protocol defined doses.
  Interventions: Drug: INCB161734; Drug: Rifampin
- Cohort 3 (Experimental): INCB161734 and esomeprazole will be administered at protocol defined doses.
  Interventions: Drug: INCB161734; Drug: Esomeprazole
- Cohort 4 (Experimental): INCB161734 and famotidine will be administered at protocol defined doses.
  Interventions: Drug: INCB161734; Drug: Famotidine

INTERVENTIONS:
Drug: INCB161734 — Oral; Tablet
Drug: Itraconazole — Oral; Tablet
  Arms: Cohort 1
Drug: Rifampin — Oral; Tablet
  Arms: Cohort 2
Drug: Esomeprazole — Oral; Tablet
  Arms: Cohort 3
Drug: Famotidine — Oral; Tablet
  Arms: Cohort 4

SUMMARY:
This study is conducted to assess the effect of itraconazole, rifampin, and acid-reducing agents on INCB161734 pharmacokinetics when administered orally in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend and willingness to sign a written ICF for the study.
* Age 18 to 55 years, inclusive, at the time of signing the ICF.
* Body mass index between 18.0 and 32.0 kg/m2 (inclusive).
* Willingness to adhere to study-related prohibitions, restrictions, and procedures.
* Ability to swallow and retain PO medication.
* Willingness to avoid pregnancy or fathering children based on the criteria defined in the prootcol.

Exclusion Criteria:

* History of uncontrolled or unstable cardiovascular, respiratory, renal, gastrointestinal, endocrine, hematopoietic, psychiatric, and/or neurological disease within 6 months of screening.
* History of rheumatologic/autoimmune disorders and immune deficiency/immunologic defects.
* History of major bleeding or thrombosis, including myocardial infarction/stroke and pulmonary embolism/deep vein thrombosis.
* Known tuberculosis infection that is active or participant-reported history of tuberculosis or treatment thereof.
* Resting pulse < 40 bpm or > 100 bpm, confirmed by repeat testing at screening.
* Presence of a malabsorption syndrome possibly affecting drug absorption (eg, Crohn disease or chronic pancreatitis).
* Any major surgery within 12 weeks of screening.
* Positive test for hepatitis B virus, hepatitis C virus, or HIV. Note: Participants whose results are compatible with prior immunization or immunity due to infection for hepatitis B may be included at the discretion of the investigator.
* Positive urine or breath test for ethanol or positive urine or serum screen for drugs of abuse that are not otherwise explained by permitted concomitant medications or diet.
* Use of tobacco- or nicotine-containing products within 1 month of screening.
* Women who are pregnant or breastfeeding.
* eGFR < 90 mL/min/1.73 m2 based on the CKD-EPI equation.
* Any history of hypersensitivity or intolerance to itraconazole, rifampin, esomeprazole or any other PPI, or famotidine or any other H2 antagonist.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2025-07-16 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics Parameter (PK): Cmax of INCB161734 | Up to 2 months
  Defined as maximum observed plasma or serum concentration of INCB161734.
Pharmacokinetics Parameter: AUC(0-t) of INCB161734 | Up to 2 months
  Defined as the area under the concentration-time curve up to the last measurable concentration of INCB161734.
Pharmacokinetics Parameter: AUC 0-∞ of INCB161734 | Up to 2 months
  Defined as the area under the concentration-time curve from 0 to infinity of INCB161734.

SECONDARY OUTCOMES:
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to 2 months
  Defined as adverse events reported for the first time or the worsening of a pre-existing event, occurring after first dose of study drug.
Pharmacokinetics Parameter: Tmax of INCB161734 | Up to 2 months
  Defined as the time to reach the maximum plasma concentration of INCB161734.
Pharmacokinetics Parameter: t1/2 of INCB161734 | Up to 2 months
  Defined as the apparent terminal phase disposition half-life of INCB161734.
Pharmacokinetics Parameter: CL/V of INCB161734 | Up to 2 months
  Defined as the apparent oral dose clearance of INCB161734.
Pharmacokinetics Parameter: Vz/F of INCB161734 | Up to 2 months
  Defined as the apparent oral dose volume of distribution of INCB161734.
Pharmacokinetics Parameter: AUC%extrap of INCB161734 | Up to 2 months
  Defined as percentage of AUC∞ (_obs, _pred) due to extrapolation from time of last measurable observed concentration to infinity of INCB161734.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (1):
- Fortrea Clinical Research Unit Ltd Labcorp Clinical Research Unit Limited Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A study to Assess the Effect of Itraconazole, Rifampin, and Acid-Reducing Agents on INCB161734 Pharmacokinetics When Administered Orally in Healthy Participants — https://www.incyteclinicaltrials.com/trials/INCB161734-103